CLINICAL TRIAL: NCT00111371
Title: Dopaminergic Enhancement of Learning and Memory (LL_001, Project on Dyslexia)
Brief Title: Dopaminergic Enhancement of Learning and Memory in Healthy Adults and Patients With Dyslexia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LL-001; Project on Dyslexia
Record Dates: First submitted 2005-05-19; First posted 2005-05-20 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2006-09

CONDITIONS: Dyslexia
Keywords: artificial grammar learning; dyslexia; healthy subjects; levodopa; drug; treatment; intervention
MeSH Terms: conditions — Dyslexia | interventions — Levodopa

INTERVENTIONS:
Drug: Levodopa

SUMMARY:
This study aims to determine whether levodopa, in combination with a high frequency training of (grammatical) rules, is effective in boosting learning success in healthy subjects and whether this kind of training in combination with levodopa improves reading and spelling abilities of patients with dyslexia.

DETAILED DESCRIPTION:
Prior work by our group shows that d-amphetamine and the dopamine precursor levodopa markedly improve word learning success in healthy subjects. In this randomized, placebo-controlled, double-blind trial, we probe whether daily administration of levodopa, coupled with a training of grammatical rules, improves the training success in healthy adults as compared to placebo administration. In the second step of this study, patients with dyslexia will be trained with the identical protocol. We postulate that the combination of intensive training in language rules and levodopa improves the reading, writing, and spelling abilities of patients with dyslexia.

ELIGIBILITY:
Inclusion Criteria:

* Right-handedness
* Age between 18-35 years
* Primary language: German

Exclusion Criteria:

* Known allergy to levodopa or tetrazine
* History of medication/drug abuse
* Acute nicotine withdrawal or > 10 cigarettes per day
* >6 cups/glasses of coffee, caffeine drinks or energy drinks per day
* >50 grams of alcohol per day
* Hypertonia
* Arteriosclerosis
* Diabetes, asthma, or glaucoma
* Psychiatric disease
* Neurologic disease
* Other medication

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-01; Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Boost in training success (percent correct) through levodopa as compared to placebo
Boost in training success (reaction times) through levodopa as compared to placebo
Increased performance on reading, spelling and writing tests in dyslexic patients treated with levodopa as compared to placebo

SECONDARY OUTCOMES:
Stability of improvements one month post training

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Knecht, Prof. Dr., Principal Investigator — Dept. of Neurology, Universityclinic of Muenster
Locations (1):
- Dept. of Neurology, University Hospital of Muenster, Münster, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Knecht S, Breitenstein C, Bushuven S, Wailke S, Kamping S, Floel A, Zwitserlood P, Ringelstein EB. Levodopa: faster and better word learning in normal humans. Ann Neurol. 2004 Jul;56(1):20-6. doi: 10.1002/ana.20125. PMID 15236398
- [Background] Breitenstein C, Knecht S. [Language acquisition and statistical learning]. Nervenarzt. 2003 Feb;74(2):133-43. doi: 10.1007/s00115-002-1466-1. German. PMID 12596014
- [Background] Opitz B, Friederici AD. Brain correlates of language learning: the neuronal dissociation of rule-based versus similarity-based learning. J Neurosci. 2004 Sep 29;24(39):8436-40. doi: 10.1523/JNEUROSCI.2220-04.2004. PMID 15456816